CLINICAL TRIAL: NCT02146300
Title: Effect of the Nasal Provocation on the Breathing Style and on the Calibration of Respiratory Effort Belts
Brief Title: Effect of the Nasal Provocation on the Breathing Style
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Oulu University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Diary number 15/2014
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Birch Pollen Allergy; Healthy Control Subjects
Keywords: birch pollen; allergy; breathing; pattern; exposure
MeSH Terms: conditions — Hypersensitivity; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Allergen and xylometatsolin (Experimental): Two separate exposure sessions: 1) nasal birch pollen exposure 2) nasal xylometazoline exposure
  Interventions: Biological: 1. session birch pollen nasal exposure 2. session xylometazoline nasal exposure

INTERVENTIONS:
Biological: 1. session birch pollen nasal exposure 2. session xylometazoline nasal exposure — Aquagen SQ 10 000 SQ/ml nasal exposure Xylometazoline 1 mg/ml nasal exposure

SUMMARY:
The purpose of this study is to find out how the provocation of the nose changes breathing style (specifically, frequency and tidal volume changes)

DETAILED DESCRIPTION:
It is intended to clarify on both healthy and birch pollen allergic adults how the provocation of the nose with the birch pollen, dilutant and xylometazoline affect the breathing style (breathing pattern) and how these possible changes could be controlled in the measurement of the breathing with respiratory effort belts. In addition to this, our intention is to clarify the effect of the facial mask on the breathing.

The allergic and control subjects undergo nasal provocation in 2 sessions. The first is done with birch pollen extract (should block the nose in allergic subjects) and the second with xylometazoline (should open the nose).

The mask group undergo similar measurements without nasal exposures.

The second objective of the study is to clarify if there are differences between the allergic and control subjects in the function of the autonomous nervous system during these provocations. This is done with the heart rate variability analysis method.

ELIGIBILITY:
Inclusion Criteria:

* Birch pollen allergic subjects must have clear nasal symptoms during the birch pollen season and birch specific IgE >= 0.70
* Healthy subjects: birch specific IgE < 0.35
* The subjects are not allowed to be under medication that affects the function of their nose during a specific time period before the measurement
* They have to be free of any acute respiratory symptoms during the prior two weeks to the measurements
* Before measurement, they are not allowed to have heavy meal or sport
* They are not allowed to have caffeine or other stimulants for 12 hours or alcohol for 24 hours.

Exclusion Criteria:

* Heart diseases
* Brain circulatory disorders
* Surgical operations of nose
* Chronic nasal symptoms
* Pregnancy
* Smoker

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
breathing style | continuously during 2 hours
  frequence and volume of breathing measured with spirometry and respiratory effort belts

SECONDARY OUTCOMES:
thorax - abdomen relation | continuously during 2 hours
  relation of the movements of the thorax and abdomen as measured with the respiratory belts
activation of the autonomous nervous system | continuously during 2 hours
  activity of the autonomous nervous system as measured with heart rate variability

CONTACTS AND LOCATIONS:
Overall Officials: Tiina M Seppänen, PhD, Principal Investigator — University of Oulu; Miia-Liisa Vakkuri, Med Cand, Principal Investigator — University of Oulu; Tapio Seppänen, Prof, Study Chair — University of Oulu; Olli-Pekka Alho, Prof, Study Chair — University of Oulu
Locations (1):
- Oulu University hospital, dept of Otorhinolaryngology, Oulu, Oulu, Finland